CLINICAL TRIAL: NCT02209220
Title: Impact of Automatic Positive Airway Pressure on Treatment Compliance in Obstructive Sleep Apnea Patients Awaiting Bariatric Surgery
Brief Title: Impact of Automatic Positive Airway Pressure on Treatment Compliance in OSA Patients Awaiting Bariatric Surgery
Acronym: APAP-CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: GROUPE DE RECHERCHE EN SANTÉ RESPIRATOIRE DE L'UNIVERSITÉ LAVAL (GESER) (Unknown)
Responsible Party: Principal Investigator, Frédéric Sériès, Principal investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APAP-21014
Record Dates: First submitted 2014-06-25; First posted 2014-08-05 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Obstructive Sleep Apnea; Treatment Compliance; Automatic Positive Airway Pressure
Keywords: Obstructive sleep apnea; Treatment compliance; Automatic positive airway pressure; Continuous positive airway pressure; Bariatric surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automatic positive airway pressure (Active Comparator): Automatic positive airway pressure treatment of obstructive sleep apnea
  Interventions: Device: Positive airway pressure for the treatment of OSA
- Continuous positive airway pressure (Active Comparator): Continuous positive airway pressure for the treatment of obstructive sleep apnea
  Interventions: Device: Positive airway pressure for the treatment of OSA

INTERVENTIONS:
Device: Positive airway pressure for the treatment of OSA
  Other Names: Positive pressure device used: ResMed Autoset S9.

SUMMARY:
Obstructive sleep apnea (OSA) is a syndrome characterized by intermittent dynamic obstruction of the upper airways that causes a fall in oxygen saturation, reflex sympathetic activation and sleep micro-arousals. In surgical patients, OSA is a well-known risk factor for perioperative complications. At Institut Universitaire de cardiologie et de Pneumologie de Quebec (IUCPQ), the investigators perform more than 450 bariatric surgeries per year. Consequently, the identification and management of OSA in this high-risk surgical population is an essential part of practice. Actual guidelines recommend that treatment for OSA be initiated before the surgical procedure. Presently, the first line treatment for OSA is continuous positive airway pressure (CPAP) therapy delivering a fixed pressure continuously to maintain the patency of the upper airways. However the compliance to this therapy is poor. An available alternative is automatic positive airway pressure (APAP) which delivers a variable amount of pressure to prevent reduction in airflow that accompanies upper airway obstruction. The APAP delivers the lowest pressure needed to prevent upper airways collapse. APAP significantly reduces the mean level of pressure delivered in comparison to conventional treatment. Theoretically, it seems logical that applying the lowest pressure necessary would allow a better device-patient synchrony and therefore improve patient's comfort.Recent trials comparing APAP and CPAP have shown that APAP is non-inferior to CPAP in controlling obstructive events. APAP would be a valuable alternative if it was not for its excess cost. However, APAP improves compliance to treatment in two types of population: poor compliant subjects and those needing high pressure levels. The investigators know that compliance to positive pressure is poor in patients without excessive daytime sleepiness, which represents the majority of patient waiting bariatric surgery. Moreover, in patients needing levels of pressure ≥ 10 water cm (cmH20), APAP improves treatment compliance, minimises side effects and improves quality of life. The review of 180 files of OSA patients treated by CPAP who had bariatric surgery in our center in 2012 demonstrated that the majority of patients needed high level pressure. These values suggest that APAP could improve treatment compliance in apneic patients waiting for bariatric surgery because they are usually poorly symptomatic and they generally require high positive pressure level.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with a BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with additional risk factors for cardiovascular disease and eligible for bariatric surgery;
* Laparoscopic bariatric surgery planned in 2-6 months. Procedures include biliopancreatic diversion with duodenal switch and sleeve gastrectomy;
* Recent diagnosis of obstructive sleep apnea made by a sleep study. The sleep study must be a overnight pulse oximetry showing a 3% desaturation index ≥ 25/hour or a polysomnography with a apnea + hypopnea index (AHI) ≥ 25/hour* ;
* No previous use of positive airway pressure device;
* ≥18 year old.

Exclusion Criteria:

* Severe comorbidities (respiratory, cardiac, neurologic or metabolic unstable disease);
* Central sleep apnea;
* Obesity hypoventilation syndrome;
* Planned bariatric surgery by laparotomy;
* Contraindications to positive airway pressure therapy: pneumothorax within the preceding 6 months, cerebrospinal fluid leak, cranial surgery or trauma within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Compliance of APAP and CPAP | at time of surgery
  Total utilisation time, daily hours of utilisation, percentage of nights with positive pressure

SECONDARY OUTCOMES:
Mean pressure level with APAP and CPAP | at time of surgery
  Pressure applied (mean pressure and 90th/95th percentile), apnea hypopnea index, amount of mask leaks.
Mean pressure level with APAP and CPAP | 1 month
  Pressure applied (mean pressure and 90th/95th percentile), apnea hypopnea index, amount of mask leaks.
Residual apnea + hypopnea index | at time of surgery
  Number of residual respiratory events recorded by the positive pressure device during the treatment period
Residual apnea + hypopnea index | 1 month
  Number of residual respiratory events recorded by the positive pressure device during the treatment period
epworth sleepiness score | at time of surgery
  Somnolence measured by Epworth Sleepiness Scale;
quality of life score with APAP and CPAP | at time of surgery
  Quality of life measured by Questionnaire sur la Qualité de vie du Québec
Positive pressure therapy adverse events | at time of surgery
  Positive airway pressure adverse effects measured by a visual analogic scale.
Compliance of APAP and CPAP | 1 month
  Total utilisation time, daily hours of utilisation, percentage of nights with positive pressure

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Séries, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Kaw R, Chung F, Pasupuleti V, Mehta J, Gay PC, Hernandez AV. Meta-analysis of the association between obstructive sleep apnoea and postoperative outcome. Br J Anaesth. 2012 Dec;109(6):897-906. doi: 10.1093/bja/aes308. Epub 2012 Sep 6. PMID 22956642
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Kuna ST, Reboussin DM, Borradaile KE, Sanders MH, Millman RP, Zammit G, Newman AB, Wadden TA, Jakicic JM, Wing RR, Pi-Sunyer FX, Foster GD; Sleep AHEAD Research Group of the Look AHEAD Research Group. Long-term effect of weight loss on obstructive sleep apnea severity in obese patients with type 2 diabetes. Sleep. 2013 May 1;36(5):641-649A. doi: 10.5665/sleep.2618. PMID 23633746
- [Background] Smith I, Lasserson TJ. Pressure modification for improving usage of continuous positive airway pressure machines in adults with obstructive sleep apnoea. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD003531. doi: 10.1002/14651858.CD003531.pub3. PMID 19821310
- [Background] Parish JM, Miller BW, Hentz JG. Autotitration positive airway pressure therapy in patients with obstructive sleep apnea who are intolerant of fixed continuous positive airway pressure. Sleep Breath. 2008 Aug;12(3):235-41. doi: 10.1007/s11325-007-0158-2. Epub 2007 Nov 28. PMID 18043955
- [Background] Wolkove N, Baltzan M, Kamel H, Dabrusin R, Palayew M. Long-term compliance with continuous positive airway pressure in patients with obstructive sleep apnea. Can Respir J. 2008 Oct;15(7):365-9. doi: 10.1155/2008/534372. PMID 18949106
- [Background] Massie CA, McArdle N, Hart RW, Schmidt-Nowara WW, Lankford A, Hudgel DW, Gordon N, Douglas NJ. Comparison between automatic and fixed positive airway pressure therapy in the home. Am J Respir Crit Care Med. 2003 Jan 1;167(1):20-3. doi: 10.1164/rccm.200201-022OC. Epub 2002 Oct 4. PMID 12406840
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Lacasse Y, Bureau MP, Series F. A new standardised and self-administered quality of life questionnaire specific to obstructive sleep apnoea. Thorax. 2004 Jun;59(6):494-9. doi: 10.1136/thx.2003.011205. PMID 15170032
- [Derived] Kermelly SB, Lajoie AC, Boucher ME, Series F. Impact of continuous positive airway pressure mode on adherence to treatment in obstructive sleep apnea patients awaiting bariatric surgery. J Sleep Res. 2021 Oct;30(5):e13288. doi: 10.1111/jsr.13288. Epub 2021 Feb 6. PMID 33547713